CLINICAL TRIAL: NCT05319522
Title: The Influence of Irisin/FNDC5 on Bone Mineral Density and Fracture Risk in Individuals With Spinal Cord Injury
Brief Title: The Relationship Between Irisin and Bone Health in Individuals With Spinal Cord Injury
Acronym: IBSCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B3641-M
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Spinal Cord Injury
Keywords: Spinal cord injuries; Irisin; Bone mineral density; Exercise
MeSH Terms: conditions — Spinal Cord Injuries; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Individuals with SCI (Active Comparator): Male and female, Veteran and non-Veteran participants with traumatic SCI will complete the baseline blood draw, muscle biopsy and DXA/HR-pQCT bone imaging. This group will complete blood draws before and after arm ergometer high-intensity interval exercise bout.
  Interventions: Behavioral: Acute Exercise
- Controls (No SCI) (Active Comparator): Male and female Veterans, age and sex-matched to participants with SCI will complete the baseline blood draw, muscle biopsy and DXA/HR-pQCT bone imaging. This group will complete blood draws before and after arm ergometer high-intensity interval exercise bout.
  Interventions: Behavioral: Acute Exercise

INTERVENTIONS:
Behavioral: Acute Exercise — Participants with and without SCI will complete an arm ergometer, high-intensity interval exercise bout. The exercise bout will be performed at a relative intensity based on previously determined peak power output during an arm ergometer graded exercise test.
  Other Names: Arm Ergometer Exercise; High-Intensity Interval Exercise

SUMMARY:
This study will examine the relationship between circulating irisin and bone health individuals with spinal cord injury. Additionally, this study seeks to examine the influence of muscle fiber type on circulating irisin and identify an exercise-based means to increase irisin concentrations.

DETAILED DESCRIPTION:
After spinal cord injury (SCI), the severe sub-lesion bone loss increases lower-limb fracture risk. In addition to mechanical loading, bone homeostasis is mediated by myokines, skeletal muscle secreted factors, including irisin. This project aims to demonstrate that irisin is a key determinant of bone mineral density in sub-lesion bone, that impaired irisin mechanisms contribute to post-SCI bone loss, and identify novel modalities to leverage the osteogenic effects of irisin to improve musculoskeletal rehabilitation strategies for individuals with SCI.

The first aim of this project seeks to determine the relationship between circulating irisin and bone mineral density (BMD) in sub-lesion bones of individuals with SCI. Past research has reported positive correlations between irisin and BMD indicating that irisin is important factor in bone homeostasis. To date, the relationship between irisin and BMD, absent mechanical loading, as seen in individuals with SCI, has not been examined. Of note, irisin increases have been demonstrated to increase bone mass in healthy mice and prevent or reduce bone loss in mouse SCI models.

The second aim of this study seeks to determine if irisin concentrations are impaired as a result of pathologic changes in sub-lesion skeletal muscle after SCI. Irisin is released into circulation following cleavage of its precursor protein which is highly expressed in skeletal muscle. Generally, healthy human muscle demonstrates a mix of type I and type II muscle fibers, however, after SCI, there is a pathological transformation from type I to type II muscle. Given that irisin's precursor protein is more highly expressed in type I muscle, the post-SCI fiber type transformation could significantly attenuate circulating irisin concentrations and impair its downstream signaling effects. Understanding whether post-SCI fiber type shifts are associated with reduced circulating irisin could help explain the inefficacy of current rehabilitation methods.

The third aim of this study seeks to measure the irisin response to arm ergometer high intensity interval exercise. If circulating irisin concentrations are important to bone health, as current research suggests, then identifying a means in increase circulating irisin is essential to developing better musculoskeletal rehabilitation methods. While exercise has been demonstrated to increase circulating irisin, the exercise modalities performed (running, whole body resistance training) are not feasible for individuals with SCI. Arm ergometry exercise could provide a means to increase circulating concentrations of this osteogenic factor.

ELIGIBILITY:
Inclusion Criteria:

Participants with SCI:

* age 18 years or older
* traumatic SCI at the cervical level 4 or lower that occurred at least 12 months prior to the start of the study
* American Spinal Injury Association Impairment Scale A, B or C
* uses a manual wheelchair as primary means of mobility (30+ hours per week)
* is able to perform a transfer independently to and from a wheelchair
* has adequate strength and upper extremity function to operate an arm ergometer

Control Participants:

* age and sex-matched to participant with SCI

Exclusion Criteria:

Participants with SCI:

* active use of medications which potentially affect bone metabolism, including: parathyroid hormone and analogs, androgenic or estrogenic steroids, bisphosphonates, oral glucocorticoids (use for more than 3 months)
* history of fractures or dislocations in the upper extremity from which the participant has not fully recovered
* upper limb pain or injury that interferes with the ability to perform aerobic exercise
* recent hospitalization for any reason (within the past three months)
* history of coronary artery disease, coronary bypass surgery or other cardiorespiratory events or conditions
* likely to experience clinically significant autonomic dysreflexia and/ or orthostatic hypotension in response to vigorous exercise
* endocrinopathy or metabolic disorders of the bone

  * e.g. Paget's disease, renal bone disease
* history of allergic reaction to lidocaine
* any other conditions that the person's primary care physician deems is a contraindication to participation in arm ergometry exercise stress testing or vigorous exercise
* pregnant
* participation in another "Greater than Minimal Risk" study.

Control Participants:

* active use of medications which potentially affect bone metabolism, including: parathyroid hormone and analogs, androgenic or estrogenic steroids, bisphosphonates, oral glucocorticoids (use for more than 3 months)
* history of neuromuscular conditions which could influence muscle gene expression
* history of lower body musculoskeletal injuries from which the participant has not fully recovered
* recent hospitalization for any reason (within the past three months)
* history of allergic reaction to lidocaine
* any other conditions that the person's primary care physician deems is a contraindication to the performance of a vastus lateralis muscle biopsy
* pregnant
* participation in another "Greater than Minimal Risk" study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Irisin - Bone measure correlations | Baseline; at rest
  Circulating irisin concentrations will be correlated with DXA and HR-pQCT bone measures
FNDC5 gene expression | Baseline; at rest
  FNDC5 gene expression will be measured in vastus lateralis skeletal muscle biopsies via RT-PCR to determine if potential differences in circulating irisin concentrations may be attributed to differential gene expression.
Exercise induced change in irisin concentration | baseline and immediately post-exercise
  Circulating irisin concentrations will be measured before and immediately following an arm ergometer high-intensity interval exercise bout to determine if this exercise modality can increased circulating irisin concentrations in individuals with SCI and controls

CONTACTS AND LOCATIONS:
Overall Officials: Adam J. Sterczala, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-11-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT05319522/ICF_000.pdf